CLINICAL TRIAL: NCT03336918
Title: Lithium Effects on the Brain's Functional and Structural Connectome in the Treatment of Bipolar Disorder
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Amit Anand, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 17-441
Record Dates: First submitted 2017-10-05; First posted 2017-11-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder; Bipolar I Depression; Bipolar II Depression; Bipolar Depression; Depression; Major Depressive Episode
Keywords: Bipolar Disorder; Bipolar I and II Depression; Lithium; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lithium; Lithium Carbonate; Citric Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gene Expression RNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Bipolar Disorder I or II Depressed: DSM-V Bipolar I or II Depressed treated with lithium
  Interventions: Drug: Lithium
- Healthy Controls: Healthy Controls with no psychiatric history

INTERVENTIONS:
Drug: Lithium — Open-label lithium treatment for Bipolar Disorder Subjects
  Healthy Controls only repeat testing - no intervention
  Other Names: Lithium carbonate or citrate or Lithium extended release
  Groups: Bipolar Disorder I or II Depressed

SUMMARY:
Lithium is highly effective in the treatment of bipolar disorder. This study aims to investigate, for the first time, the impact of lithium monotherapy on the structural and functional connectivity of the brain using MRI imaging.

DETAILED DESCRIPTION:
The premise of this proposal is that the clinical efficacy of lithium in bipolar disorder, and its complex effects on multiple brain physiological functions, may be best deciphered using a network properties-metric approach. This approach is critical because it provides insight into the function of brain networks (e.g., resilience to disruption, central hubs), which is likely to be more closely linked to behavioral outcomes. Furthermore, we will conduct an exploratory investigation of the in vivo molecular effects of lithium by measuring peripheral gene expression. To bring these together, we will also explore whether connectome changes serve as mediator between molecular changes (i.e., gene expression) induced by lithium treatment and behavioral changes (e.g., depression, mood stability, suicidality).

ELIGIBILITY:
Inclusion criteria for BD subjects:

* ages 18-60 years (inclusive) and able to give voluntary informed consent;
* Satisfy criteria for Diagnostic and Statistical Manual 5th edition (DSM-V) for BD I or II, current Depressive Episode;
* 17-item Hamilton Depression Rating Scale (HAM-D) score >15 and <25;
* Young Mania Rating Scale (YMRS) < 8;
* no psychotropics in the last 2 weeks (if previously on fluoxetine then medication free for 5 weeks) OR on stable psychotropic medications for 12 weeks
* no lithium treatment for past 6 months;
* satisfy criteria to undergo an MRI scan based on MRI screening questionnaire;
* able to be managed as outpatients during the study as ascertained by Clinical Global Severity Scale < 5 (i.e., moderately ill) and no significant suicidal or homicidal ideation or gross disability.

Exclusion criteria for BD subjects are:

* meeting DSM-IV criteria for schizophrenia, schizoaffective disorder, or an anxiety disorder as
* a primary diagnosis;
* requiring inpatient treatment;
* meeting DSM-V criteria for substance dependence within the past 3 months, except caffeine or nicotine;
* positive urinary toxicology screening at screening visit;
* use of alcohol in the past 1 week;
* serious medical or neurological illness;
* current pregnancy or breast feeding;
* metallic implants or other contraindications to MRI.

Inclusion criteria for healthy subjects:

* ages 18-60 years and ability to give voluntary informed consent;
* no history of psychiatric illness or substance abuse or dependence;
* no significant family history of psychiatric or neurological illness in first degree relative;
* not currently taking any prescription or centrally acting medications;
* no use of alcohol in the past 1 week;
* and no serious medical or neurological illness.

Exclusion criteria for healthy subjects are:

* under 18 years of age;
* pregnant or breast-feeding;
* metallic implants or other contraindication to MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Bipolar disorder and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity (Fc) changes | 2, 8, 26 weeks
  Investigate effects of lithium monotherapy treatment of BD on changes in Fc through fMRI imaging from baseline after 2, 8, and 26 weeks of treatment and test whether these changes correlate with improvement in state-related symptoms and longer term mood stability. Healthy controls will also be scanned at the same time points but not treated.
Structural Connectivity (Sc) changes | 2, 8, 26 weeks
  Investigate effects of lithium monotherapy treatment of BD depression on changes in the diffusion weighted imaging Sc through fMRI imaging from baseline after 2, 8, and 26 weeks and test whether these changes correlate with depression severity and mood stability. Healthy controls will also be scanned at the same time points but not treated.

SECONDARY OUTCOMES:
Changes in peripheral gene expression | 2, 8, 26 weeks
  An exploratory investigation of whether lithium-related changes in the functional and structural connectome over time represent a link between shifts in peripheral gene expression and improvement in illness-related measures.Lithium therapy will be associated with changes in gene expression pathways such as the mitochondrial-carnitine shuttle pathway, which in turn will be related to changes in the functional and structural connectome.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation Center for Behavioral Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided